CLINICAL TRIAL: NCT01596946
Title: Home-sampling as a Tool in a Chlamydia Trachomatis Partner Notification Context. A Multi-centre Cluster-randomized Controlled Trial.
Brief Title: Home-sampling in Partner Notification of Chlamydia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostergotland County Council, Sweden (Other)
Collaborators: Medical Research Council of Southeast Sweden (Other Government)
Responsible Party: Principal Investigator, Lars Falk, MD PhD consultant, Ostergotland County Council, Sweden
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: Forss8743, LiO 201 261
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Chlamydia
Keywords: contact tracing; home sampling; cluster randomisation
MeSH Terms: conditions — Chlamydia Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contact tracing mode test at clinic (Active Comparator): Conventional mode of contact tracing where the partners were asked by either the index patient or demanded by the counsellor to attend a clinic for C. trachomatis testing. The date of testing for chlamydia of the study subject i e a sexual partner to a chlamydia infected index patient was noted. Those partners being C trachomatis positive were referred to the STD-clinic for contact tracing and following the same study arm a the index patient.
  Interventions: Behavioral: Contact tracing mode test at clinic
- Self-sampling at home (Experimental): The intervention: Self-sampling of sexual partners to infected index patient for chlamydia by urine test or vaginal sampling at home. They sent the kit tube to a microbiological laboratorium for analysis. The test kit was sent by post by the counsellor at the STD-clinic or distributed via the index patient. The partner in this arm was informed about the test result from the STD-clinic and those tested C trachomatis positive were given an appointment for treating and contact tracing as soon as possible. Their partners were not randomised but following the same mode. The days from the counselling conversation with the index patient to the date of testing was measured and compared with partners tested following arm 1 mode.
  Interventions: Behavioral: Self-sampling at home - Sent Test Kit

INTERVENTIONS:
Behavioral: Contact tracing mode test at clinic
  Arms: Contact tracing mode test at clinic
Behavioral: Self-sampling at home - Sent Test Kit
  Arms: Self-sampling at home

SUMMARY:
Though partner notification is mandatory to perform of Chlamydia trachomatis infected individuals in Sweden, there was a 10-15% annually increase of reported cases between 1997 and 2007 indicating that partner notification may not be effective in preventing transmission. The investigators wanted to determine whether there was any difference in time between home-sampling and clinical testing as a tool of partner notification measured from eliciting of partners to date of testing.

ELIGIBILITY:
Inclusion Criteria:

* Sexual Partners to chlamydia infected index patients accepting to participate in the study.

Exclusion Criteria:

Index patients not living in Sweden or not speaking Swedish.

* MSM.
* Sexual partners living in another county or abroad.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 633 (Actual)
Dates: Start 2006-11; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Difference in time, measured as days from the meeting between the index patient and the counsellor (i.e. the eliciting of sexually partners) until the date of C. trachomatis testing of partners | 60 days or more were defined as an exclusion criterion
  Difference in time, measured as days from the meeting between the index patient and the counsellor (i.e. the eliciting of sexually partners) until the date of C. trachomatis testing of partners, if sexual partners had attended a clinic for testing or had the opportunity of home-sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Falk, MD PhD, Principal Investigator — Östergötland CC
Locations (1):
- R&D department of Local Health Care, Linköping, Sweden